CLINICAL TRIAL: NCT04192162
Title: Effects of Sulfur Water and Mud Therapy on Serotonin Activity and Biochemical Parameters in Patients' Osteoarthrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Specialized Rehabilitation Hospital Banja Koviljaca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRH BanjaKoviljaca
Record Dates: First submitted 2019-11-12; First posted 2019-12-10 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis of Multiple Joints
Keywords: osteoarthritis; balneotherapy; mud therapy; sulfuric water; serotonin
MeSH Terms: conditions — Osteoarthritis | interventions — Mud Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of sulfur balneotherapy and mud pack therapy (Experimental): Experimental group patients underwent sulfur balneotherapy and mud pack therapy. The duration of spa therapy program was 12 days.From the blood of patients, serotonin values, parameters of complete blood count, lipid status and inflammatory markers were analyzed before and after the therapy.
  Interventions: Other: Mud therapy application; Other: Sulfur water application
- Group of sulfur balneotherapy, mud pack therapy and exercise (Active Comparator): Control group of patients had mud pack therapy, sulfur balneotherapy and exercise in hygienic water. This group is a hydro group. From the blood of patients we analyzed parameters od complete blood count, serotonin values, lipid status and inflammatory markers before and after the therapy.
  Interventions: Other: Mud therapy application; Other: Sulfur water application; Other: Hygienic water

INTERVENTIONS:
Other: Mud therapy application — Aplication the mud pack therapy from 20 minutes
  Other Names: mud pack
Other: Sulfur water application — Aplication the sulfur water in bath from 20 minutes
  Other Names: Sulfur bath
Other: Hygienic water — Exercise in hygienic water
  Other Names: Exercise in hygienic water
  Arms: Group of sulfur balneotherapy, mud pack therapy and exercise

SUMMARY:
This study is to examine the effects of sulfur bath and mud therapy on serotonin levels and other biochemical parameters in the blood of the osteoarthritis patients, as well as water the application of exercise in water effects the results we receive.

DETAILED DESCRIPTION:
Sulfur baths and mud packs are known to have a positive effect in patients with osteoarthritis (OA). OA is a chronic degenerative disease accompanied by a constant pain that often leads to changes in the mood of patients. Over the last few decades, numerous articles reported various beneficial effects of sulfur water and peloid therapeutic applications. Serotonin is one of the important neurotransmitters that have numerous functions such as regulation of body temperature, sleep, appetite, while its main function is reflected in controling of depression.

The aim of this study is to examine the effects of sulfur bath and mud therapy on serotonin levels and other biochemical parameters in the blood of the OA patients, as well as whether the application of exercise in water effects the results we receive.

Randomized controlled study included patients with hip and/or knee OA both sexes, randomized into two groups. The first group patients underwent sulfur balneotherapy and mud pack therapy. Patients in the second group had sulfur balneotherapy, mud pack therapy and exercise in hygienic water. The duration of spa therapy program was 12 days. Serotonin values, parameters of complete blood count, lipid status and inflammatory markers were analyzed before and after the therapy.

This study is expected to be another contribution to existing evidence and shed light on the mechanisms of beneficial effects of balneotherapy and mud therapy and whether addition underwater exercise would have extra therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

1. Ages of 50 - 65 , both sexes
2. Patients diagnosed with hip and / or knee OA without having used balneotherapy in the previous year
3. Patients who have not changed their medication in the last 2 months
4. Patients who have not received injections into the hip and / or knee joint in the last 6 months (PRP, Diprofos…)

Exclusion Criteria:

1. Secondary hip and / or knee OA
2. Patients with MOA inhibitors, selective serotonin inhibitors, morphine, lithium and methyldopa in therapy
3. Visible disruption of hip and / or knee joint structures
4. Treatment of malignancy
5. Diseases of the heart, lungs, decompensated conditions of other organs, infections, active bleeding
6. Severe hip and / or knee joint injuries, fractures, and previous surgical procedures
7. Physical therapy, balneotherapy back one year

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-04-18 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
The serotonin levels | Time Frame: Baseline vs. 12-days
  Serotonin concentration

SECONDARY OUTCOMES:
Marker of inflammation | Time Frame: Baseline vs. 12-days
  Sedimentation concentration
Analysis of hemoglobin | Time Frame: Baseline vs. 12-days
  Concentration of hemoglobin (g/L)
Analysis of red blood cell counts | Time Frame: Baseline vs. 12-days
  The total number of erythrocytes / L

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar M Jokić, Principal Investigator — Specijalna bolnica za rehabilitaciju Banja Koviljača
Locations (1):
- Specializd Rehabilitation Hospital Banja Koviljaca, Loznica, Banja Koviljaca, Serbia

IPD SHARING:
Plan to Share IPD: No